CLINICAL TRIAL: NCT01703676
Title: Klinefelter Syndrome: Do the Parental Origin and Epigenetic Profile of the Supernumerary X Chromosome Determine Phenotype, Morbidity, Inflammatory Status and Cardiovascular Risk?
Brief Title: Epigenetics and Metabolic Disorders in Men With the Klinefelter Syndrome
Acronym: IZKF-CRA03-09
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Zitzmann, Clinical Andrology, University Hospital Muenster
Other Study IDs: EpigenMetabDisordKlinefelter
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Klinefelter Syndrome, Hypogonadism
Keywords: Hypogonadism, Klinefelter Syndrome, Cardiovascular Risk, Epigenetics, Methylation of Genes; Cardiovascular risk factors; Gonadal status; Gene expression; Methylation
MeSH Terms: conditions — Klinefelter Syndrome; Hypogonadism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Testicular Tissue, Mouth Epithelium
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Patients: Klinefelter Patients
- Parents: Parents of Klinefelter Patients
- Controls M: Healthy Male Control with normal karyotype
- Controls F: Healthy female controls

SUMMARY:
This study will elucidate how the parental origin of the X-chromosome influences health status as well as metabolic fate in Klinefelter patients. Epigenetics and transcriptome-research will be directly linked to the metabolic and inflammatory pattern of actual patients to improve care for them. The Klinefelter Syndrome is one of the most common genetic disorders in men. The patients have one supernumerary X-chromosome, which is partly active and disturbs a normal male development. Testosterone deficiency in form of primary hypogonadism is a common feature in these men. Such a condition promotes clinically relevant metabolic patterns related to a pro-inflammatory status and diabetes mellitus type 2 (insulin resis-tance), cardiovascular disease as well as infertility. However, the variety of pathologies is pro-nounced between patients and low testosterone concentrations cannot fully explain the wide scope of pathologies in these men. Some patients become clinically obvious during puberty and adoles-cence, some in their thirties or later and all exhibit a huge variation in phenotype. Switching on and off of specific genes on the X-chromosome is differential, depending on the origin either from the maternal or paternal side. Hence, an influence on the clinical picture is hypothesised. Thus, key targets are clarification of the parental origin of the supernumerary X chromosome and elucidation of methylation and expression profile of pivotal X-chromosomal genes. These will be related to clinically relevant metabolic and inflammatory patterns as well as fertility to identify individual risks as well as treatment strategies for Klinefelter patients.

ELIGIBILITY:
Inclusion Criteria:

Klinefelter Syndrome

Exclusion Criteria:

Mosaic status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients, their parents, male controls, female controls
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zitzmann, MD, PhD, Principal Investigator — University Hospital Muenster

REFERENCES:
- [Derived] Zitzmann M, Bongers R, Werler S, Bogdanova N, Wistuba J, Kliesch S, Gromoll J, Tuttelmann F. Gene expression patterns in relation to the clinical phenotype in Klinefelter syndrome. J Clin Endocrinol Metab. 2015 Mar;100(3):E518-23. doi: 10.1210/jc.2014-2780. Epub 2014 Dec 22. PMID 25532039